CLINICAL TRIAL: NCT04809246
Title: Prisons Evaluation of a One-stop-shop InterVentiOn to Scale-up Hepatitis C Testing and Treatment (PIVOT)
Brief Title: Prisons Evaluation of a One-stop-shop InterVentiOn
Acronym: PIVOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kirby Institute (Other Government)
Collaborators: Justice Health & Forensic Mental Health Network NSW Australia (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: VISP0105
Record Dates: First submitted 2021-02-02; First posted 2021-03-22 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2022-01

CONDITIONS: Hepatitis C
Keywords: Hepatitis C; Public Health; Health Service; Prisons
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Intervention Model Description: This study will be conducted as a prospective historically controlled study with a primary objective of assessing the effect of an intervention integrating point-of-care HCV RNA testing, non-invasive liver fibrosis assessment, fast-tracked DAA therapy, and linkage to hepatitis care (a 'one-stop-shop' intervention) on the proportion of participants initiating DAA therapy among people who are recently incarcerated within reception correctional centre(s) in Australia.
  All people who are newly incarcerated (in the previous six weeks) will be offered participation. The first 240 individuals will be enrolled into a control period to receive HCV testing and treatment via the standard of care with the current health service model. After the control period, the next 300 individuals will be enrolled in the intervention period to receive HCV testing and treatment via the 'one-stop-shop' intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of care (No Intervention): The first group (n=240) of participants enrolled in the study will be assigned to the control period to receive the standard of care.
- 'One-stop-shop' intervention (Experimental): Following the control period, the second group (n=300) of participants enrolled in the study will be assigned to the intervention period to receive the 'one-stop-shop' intervention.
  Interventions: Other: 'One-stop-shop' hepatitis clinic

INTERVENTIONS:
Other: 'One-stop-shop' hepatitis clinic — Establishment of a 'one-stop-shop' hepatitis clinic, integrating point-of-care HCV RNA testing, followed by clinical assessment, non-invasive liver fibrosis assessment by fibro-elastography (Fibroscan), and early DAA prescription (for those with chronic HCV) followed by linkage to ongoing hepatitis care, all in the same 60-minute visit.
  Arms: 'One-stop-shop' intervention

SUMMARY:
A prospective historically controlled study to assess the effect of an intervention integrating point-of-care hepatitis C (HCV) RNA testing, non-invasive liver fibrosis assessment, fast-tracked direct-acting antiviral (DAA) prescription, and linkage to hepatitis care (a 'one-stop-shop' intervention), on the proportion of participants initiating DAA therapy among people who are recently incarcerated within reception correctional centre(s) in Australia.

ELIGIBILITY:
Inclusion criteria

1. has provided written, informed consent to participate;
2. is male and ≥18 years of age on enrolment;
3. has been incarcerated within the last six weeks;
4. is HCV DAA treatment naïve;
5. is able and willing to provide informed consent and abide by the requirements of the study.

   For HCV RNA positive participants commencing treatment:
6. if HIV-1 infected must also meet the following criteria:

   1. HIV infection documented by any licensed rapid HIV test or HIV enzyme or chemiluminescence immunoassay (E/CIA) test kit at any time prior to study entry (Baseline) and confirmed by a licensed Western blot or a second antibody test by a method other than the initial rapid HIV and/or E/CIA, or by HIV-1 p24 antigen, or plasma HIV-1 RNA viral load; and
   2. be on HIV antiretroviral therapy (ART) for at least 4 weeks prior to study entry using an ART regimen that is allowable with the selected DAA regimen as determined by the current PI and the Liverpool drug interaction website (http://www.hiv-druginteractions.org/ )

Exclusion criteria

For HCV RNA positive participants commencing treatment, the subject will be excluded if they have:

1. untreated HIV co-infection;
2. chronic HBV co-infection;
3. any clinically significant condition, history or concomitant medication known to contraindicate DAA therapy or would not be suitable for management within a prison-based treatment setting;
4. is unable to gain an accurate reading on the fibroscan or the result is invalid;
5. known clinical or laboratory evidence of cirrhosis, or cirrhosis documented on fibro-elastography (> 12.5 Kpa).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 541 (Actual)
Dates: Start 2019-10-31 (Actual); Primary Completion 2021-04-23 (Actual); Study Completion 2021-09-10 (Actual)

PRIMARY OUTCOMES:
The proportion of people who have initiated DAA therapy within 12 weeks from enrolment | 12 weeks from enrolment

SECONDARY OUTCOMES:
The proportion of people tested for HCV infection at 12 weeks from enrolment | 12 weeks from enrolment
The proportion of participants who complete DAA therapy in prison | End of Treatment (8 weeks from treatment initiation)
The proportion of people who have an end of treatment response | End of Treatment (8 weeks from treatment initiation)
The proportion of people who have an HCV treatment response (sustained virological response) | Sustained virological response at 12 weeks post treatment completion
The time taken from testing to each step in the care cascade | Varying, up to 9 months post-enrolment.
The proportion of people lost to follow-up | Varying, up to end of study (estimated to be 12 months from study commencement)
The acceptability of the 'one-stop-shop' (proportion of prisoners who refuse to participate) | Varying, up to end of subject enrolment (estimated to be 12 months from study commencement)
The proportion of people reinfected at SVR12 | Varying, up to 9 months post-enrolment.
The proportion of people reporting injecting risk behaviours (at ETR and SVR12) | Varying, up to 9 months post-enrolment.
The cost-effectiveness of the 'one-stop-shop' (cost-ratio of 'one-stop-shop' and standard of care) | End of study (estimated to be 12 months from study commencement)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Lloyd, Prof, Principal Investigator — Kirby Institute, University NSW
Locations (1):
- Mid North Coast Correctional Centre, Kempsey, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
Data may be available immediately following publication for 7 years, no end date determined, upon request to the researchers.
  Data may be available to researchers on a case-by-case basis at the discretion of Principal Investigator. Data may be available to researchers upon request for conducting IPD meta-analyses (separate ethics approval required). Access to data is subject to approvals by Principal Investigator (a.lloyd@unsw.edu.au)
Supporting Information: CSR
Time Frame: Data may be available immediately following publication for 7 years, no end date determined, upon request to the researchers.
Access Criteria: Access to data is subject to approvals by Principal Investigator (a.lloyd@unsw.edu.au). A link to the report will be provided upon publication.

REFERENCES:
- [Derived] Sheehan Y, Cunningham EB, Cochrane A, Byrne M, Brown T, McGrath C, Lafferty L, Tedla N, Dore GJ, Lloyd AR, Grebely J. A 'one-stop-shop' point-of-care hepatitis C RNA testing intervention to enhance treatment uptake in a reception prison: The PIVOT study. J Hepatol. 2023 Sep;79(3):635-644. doi: 10.1016/j.jhep.2023.04.019. Epub 2023 Apr 26. PMID 37116714
- [Derived] Lafferty L, Sheehan Y, Cochrane A, Grebely J, Lloyd AR, Treloar C. Reducing barriers to the hepatitis C care cascade in prison via point-of-care RNA testing: a qualitative exploration of men in prison using an integrated framework. Addiction. 2023 Jun;118(6):1153-1160. doi: 10.1111/add.16137. Epub 2023 Feb 12. PMID 36683132